CLINICAL TRIAL: NCT03527914
Title: Patient Generated Goals in Mental Health: Better Outcomes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Kathleen Pajer, Chief of Psychiatry, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8374
Record Dates: First submitted 2018-02-18; First posted 2018-05-17 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Mental Health
Keywords: Depression; Psychosis; Personality Disorder; Substance Abuse
MeSH Terms: conditions — Psychological Well-Being; Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Patients will receive their standard care at the Outpatient Mental Health Service
  Interventions: Other: Treatment as Usual
- Goal Based Outcomes (Experimental): Up to three goals can be tracked during treatment, although patients often decide to just focus on one. Progress on the goal is then quantitatively rated by the patient, with the provider, at every appointment. Adjustments in the care are then made in an iterative process to ensure that the goal will be met.
  Interventions: Other: Goal Based Outcomes

INTERVENTIONS:
Other: Goal Based Outcomes — Up to three goals can be tracked during treatment, although patients often decide to just focus on one. Progress on the goal is then quantitatively rated by the patient, with the provider, at every appointment. Adjustments in the care are then made in an iterative process to ensure that the goal will be met.
  Arms: Goal Based Outcomes
Other: Treatment as Usual — Patients will receive their standard care at the Outpatient Mental Health Service
  Arms: Treatment as Usual

SUMMARY:
Researchers believe that clinical care can be improved by engaging patients and families directly in planning the care process. Engagement efforts have included asking patients/families to provide information about whether they are getting better. But what does "getting better" mean? The merits of surveys, questionnaires, or rating scales have been widely discussed. Should they be disorder-specific or global? What should the investigators do if patients have difficulty reading or understanding these instruments? Investigators in the United Kingdom have proposed a simple solution: ask the patients and families what their primary goal treatment goal is and track progress together on that goal (Goal-Based Outcomes or GBO). Although there has been some work to suggest that this is helpful, it has never been tested in a controlled way. This study will do a randomized controlled trial to test whether GBO improves clinical care in child and youth mental health. Although the study will use this in child and youth mental health care, if it is successful, it can be tested and applied in any care setting with any type of medical problem. This could change practice at the Children's Hospital of Eastern Ontario (CHEO) and throughout Canada.

ELIGIBILITY:
Inclusion Criteria:

* Children and youth
* Attending outpatient mental health services at CHEO

Exclusion Criteria:

-Child and youth attending group therapy at CHEO Outpatient Mental Health Services

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 152 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Patient/Family Satisfaction | Administered at study completion (up to 52 weeks)
  Measured using the Experience of Service Questionnaire
Change in Symptoms | Administered at the first appointment and at study completion (up to 52 weeks)
  Measured using the Strengths and Difficulties Questionnaire (SDQ)
Change in Function | Administered at the first appointment and at study completion (up to 52 weeks)
  Measured using the Child Global Assessment of Functioning Scale. The total score (on a scale of 0-100) will be used, with a higher score indicating better function

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Pajer, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided